CLINICAL TRIAL: NCT04697680
Title: Efficacy of a Novel Sleep Intervention in Short Sleepers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 2020 pandemic, unable to recruit and start study
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, MICHAEL A GRANDNER, Director of Sleep and Health Research Program, Associate Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1812207442
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2021-02

CONDITIONS: Sleep
Keywords: Sleep Extension; Actigraphy; Sleep Diaries; Sleep Efficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Active Comparator): Subjects randomized into Group 1 will be provided with a sleep schedule each week based on an algorithm (Algorithm 1) calculated from sleep diaries and fitbit data. Subjects will complete questionnaires at an initial clinic visit. Subjects will then complete a sleep diary upon waking each day and wear a Fitbit Charge 2 device for sleep monitoring each day for 8 weeks. At the end of the study, subjects will complete follow-up questionnaires at a final clinic visit.
  Interventions: Behavioral: Algorithm 1
- Group 2 (Active Comparator): Subjects randomized into Group 2 will be provided with a sleep schedule each week based on an algorithm (Algorithm 2) calculated from sleep diaries and fitbit data. Subjects will complete questionnaires at an initial clinic visit. Subjects will then complete a sleep diary upon waking each day and wear a Fitbit Charge 2 device for sleep monitoring each day for 8 weeks. At the end of the study, subjects will complete follow-up questionnaires at a final clinic visit.
  Interventions: Behavioral: Algorithm 2
- Group 3 (Active Comparator): Subjects randomized into Group 1 will be provided with a sleep schedule each week based on an algorithm (Algorithm 3) calculated from sleep diaries and fitbit data. Subjects will complete questionnaires at an initial clinic visit. Subjects will then complete a sleep diary upon waking each day and wear a Fitbit Charge 2 device for sleep monitoring each day for 8 weeks. At the end of the study, subjects will complete follow-up questionnaires at a final clinic visit.
  Interventions: Behavioral: Algorithm 3

INTERVENTIONS:
Behavioral: Algorithm 1 — A sleep extension algorithm (algorithm 1) will be calculated and implemented based on information obtained from Sleep Diary and Fitbit data.
  Arms: Group 1
Behavioral: Algorithm 2 — A sleep extension algorithm (algorithm 2) will be calculated and implemented based on information obtained from Sleep Diary and Fitbit data.
  Arms: Group 2
Behavioral: Algorithm 3 — A sleep extension algorithm (algorithm 3) will be calculated and implemented based on information obtained from Sleep Diary and Fitbit data.
  Arms: Group 3

SUMMARY:
Approximately 1/3 of Americans sleep ≤6h per night, an amount that has been deemed sub-optimal by the American Academy of Sleep Medicine and Sleep Research Society, the National Sleep Foundation, American Thoracic Society, and the American Heart Association. These consensus statements echo findings from many reviews on this topic. This is alarming, given epidemiologic and experimental research showing that reduced sleep time is associated with a variety of negative health outcomes including obesity, diabetes, cardiovascular disease, and mortality. Different people may need different amounts of sleep. And some people may not be able to make large changes to their sleep schedule all at once. Many individuals have situational constraints that change over time. As such, short sleep represents an unmet public health problem. There are, however, no empirically supported interventions for insufficient sleep. The proposed study addresses this critical gap by evaluating the efficacy of a novel intervention that is theoretically grounded, feasible, and has positive impacts on sleep duration. The intervention in the proposed study is by design self-correcting, individually-tailored, and not dependent on unknown individual sleep needs. It can adapt to any schedule and situation and can adapt to changes in a person's sleep schedule. The main goal of this study is to evaluate whether a manually determined sleep extension intervention is effective at improving sleep and related outcomes among adults who find it difficult to get enough sleep.

DETAILED DESCRIPTION:
Approximately 35 % of Americans sleep ≤6h per night, an amount that has been deemed sub-optimal by the American Academy of Sleep Medicine and Sleep Research Society, the National Sleep Foundation, American Thoracic Society, and the American Heart Association. These consensus statements echo findings from many reviews on this topic. This is alarming, given epidemiologic and experimental research showing that reduced sleep time is associated with a variety of negative health outcomes including obesity, diabetes, cardiovascular disease, and mortality. As such, short sleep represents an unmet public health problem. There are, however, no empirically supported interventions for insufficient sleep. The proposed study addresses this critical gap by evaluating the efficacy of a novel intervention that is theoretically grounded, feasible, and has positive impacts on sleep duration.

Previous studies have associated habitual short sleep duration with important adverse cardiometabolic outcomes, including weight gain, obesity, diabetes, cardiovascular disease, stress, etc. They suggest that those that report short sleep may be more likely to experience functional impairments and are less likely to engage in behaviors consistent with a healthy lifestyle. A proposed mechanism of these relationships is that insufficient sleep duration triggers metabolic disturbances and increased immune response resulting in appetite dysregulation, adverse cardiovascular outcomes, and resultant disease states. In addition to cardiometabolic effects, behavioral and functional consequences of short sleep have been well-documented. For example, short sleepers are more likely to exhibit difficulties initiating and/or maintaining sleep daytime sleepiness drowsy driving, and other impairments as a result of sleep loss. Laboratory studies have extensively documented neurocognitive and behavioral effects of sleep loss, including increased objective sleepiness, impaired vigilance using computer-based psychomotor assessments, and deficits in working memory, decision-making, and executive function, as assessed using standardized neuropsychologic and neuroimaging techniques.

Most, if not all, sleep disorders have targeted interventions. Interventions have not been developed or evaluated for insufficient sleep. An effective and disseminable intervention for insufficient sleep will likely differ from those of sleep disorders- rather than an in-clinic, visit-based, medication/device/procedure-focused, non-tailored approach, a successful approach for insufficient sleep will likely be out-of-clinic, population/community-based, lifestyle-focused, and individually-tailored. The problem of insufficient sleep is less like other sleep disorders and more like other health behaviors, such as smoking, poor diet, and lack of physical activity, in that the reasons for insufficient sleep involve beliefs and attitudes, home and work demands, and environmental constraints.

With this in mind, a behavioral intervention was developed based on concepts originally implemented in Cognitive Behavioral Therapy for Insomnia (CBTI), the most well-supported treatment approach for insomnia. Although CBTI does not routinely increase sleep duration, it has sleep efficiency as its primary endpoint and employs concepts that can potentially be used to increase sleep time while maintaining high levels of sleep efficiency. The intervention originally developed included algorithms that recognize the natural "ebb and flow" of sleep ability within an individual seek to use an individual's own sleep data to predict (1) when is an optimal time to make a change to sleep, and (2) what sort of incremental change should be made with the eventual goal of increasing sleep efficiency and duration.

Different people may need different amounts of sleep. And some people may not be able to make large changes to their sleep schedule all at once. Many individuals have situational constraints that change over time. The intervention in the proposed study is by design self-correcting, individually-tailored, and not dependent on unknown individual sleep needs. It can adapt to any schedule and situation and can adapt to changes in a person's sleep schedule.

This sleep extension intervention specifically uses a novel approach, where individualized feedback will be provided to each participant, based on information provided by the wearable devices and the sleep diary. The goal is recognizing the optimal time to make a change to sleep patterns and deciding what kind of change should be made.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18-60 years old
2. Have a typical sleep schedule of <6 hours per night

Exclusion Criteria:

1. Any condition that the PI considers would significantly impede participation in the study.
2. Participant is under 18 years of age or older than 60 years of age
3. Do not have a typical sleep schedule of <6 hours per night

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep Duration | Change in sleep duration from baseline and then every 7 days, over a period of 8 weeks.
  Sleep duration will be assessed using Fitbit devices and/or sleep diaries.
Change in Sleep Efficiency | Change in sleep efficiency from baseline and then every 7 days, over a period of 8 weeks.
  Sleep efficiency will be manually calculated using information from Fitbit devices and/or sleep diaries.

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) scores across an eight (8) week study | Change from baseline and then at end of study [Day 57]
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep. In addition, a total score will be evaluated in addition to the individual items. A score of 5 has been identified as a cutoff for "poor" sleep.
Change in Insomnia Severity Index (ISI) scores across an eight (8) week study | Change from baseline and then at end of study [Day 57]
  The Insomnia Severity Index (ISI) is a brief (7-item) insomnia screening tool that is the gold standard for quantifying severity of clinical insomnia symptoms.
Change of Epworth Sleepiness Scale (ESS) scores across an eight (8) week study | Change from baseline and then at end of study [Day 57]
  ESS is a standard measure to assess daytime sleepiness and consists of 8 items ranging from "No chance of dozing" to "High chance of dozing" that evaluate sleep propensity in a range of situations.
Change in Perceived Stress Scale (PSS) scores across an eight (8) week study | Change from baseline and then at end of study [Day 57]
  The perceived Stress Scale is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. A total score is calculated for this tool.
Change in Profile of Mood States (POMS) scores across an eight (8) week study | Change from baseline and then at end of study [Day 57]
  The Profile of Mood States (POMS) is a psychological rating scale used to assess transient, distinct mood states. The POMS measures six different dimensions of mood swings over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment. A total score will be evaluated in addition to the individual items.
Change in Patient Health Questionnaire (PHQ9) scores across an eight (8) week study | Change from baseline and then at end of study [Day 57]
  PHQ9: The PHQ9 will screen for depression symptoms. It is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression: It incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool. Participants with a score >9 will be excluded. A total score is calculated for this tool.
Change in Sleep Disorders Symptom Check List (SDSCL) scores across an eight (8) week study | Change from baseline and then at end of study [Day 57]
  The SDSCL is a 20 question instrument was developed to screen for six sleep disorders (insomnia, obstructive sleep apnea, restless legs syndrome/periodic limb movement disorder, circadian rhythm sleep-wake disorders, narcolepsy, and parasomnias) and evaluated psychometrically. Answers range from "Never" to ">5 times a week".
Change in Brief Index of Sleep Control (BRISC) scores across an eight (8) week study | Change from baseline and then at end of study [Day 57]
  The BRISC is a reliable and valid screening tool to estimate self-perceived control over sleep across multiple domains. It is brief, simple, and strongly associated with overall self-reported sleep quality, insomnia, daytime sleepiness, and sleep duration. Total BRISC scores are computed as an average of item scores.
Change in Generalized Anxiety Disorder 7- Item Scale scores (GAD-7) across an eight (8) week study | Change from baseline and then at end of study [Day 57]
  The GAD-7 is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder. It contains 7 items with answers ranging from "Not at all" to "Nearly every day".
Changes in The STOP-Bang questionnaire scores across an eight (8) week study | Change from baseline and then at end of study [Day 57]
  STOP-Bang is a validated screening tool for Obstructive Sleep Apnea (OSA). The higher the STOP-Bang score, the greater is the probability of moderate-to-severe OSA.
Change in Positive and Negative Affect Scale (PANAS) across an eight (8) week study | Change from baseline and then at end of study [Day 57]
  PANAS: The Positive and Negative Affect Scales are brief screening measures that assess both positive and negative emotional experiences. This scale will allow for separate assessment of impact on both positive and negative mood.
Change in The Circadian Energy Scale (CIRENS) scores across an eight (8) week study | Change from baseline and then at end of study [Day 57]
  CIRENS is a very short and simple chronotype measurement tool based on energy. The CIRENS consists of two introspective questions about the usual energy level (very low, low, moderate, high, or very high, scored 1 to 5) in the morning and in the evening. The difference between energy level scores (-4 to 4) felt by respondents in the evening and morning defines the chronotype score and classification.
Change in the Three Factor Eating Questionnaire (TFEQ) scores across an eight (8) week study. | Change from baseline and then at end of study [Day 57]
  The Three Factor Eating Questionnaire is a validated eating behavior questionnaire that assesses eating behaviors on three subscales: cognitive restraint, emotional eating and disinhibition.
Change in Assessment of Sleep Environment (ASE) scores across an eight week study. | Change from baseline and then at end of study [Day 57]
  The ASE questionnaire is a 13 item scale which assesses difficulty sleeping due to factors of sleep environment including light, temperature, and sound, with responses ranging from "Strongly Disagree" to "Strongly Agree".
Changes in International Physical Activity Questionnaire (IPAQ) scores across an eight week study. | Change from baseline and then at end of study [Day 57]
  The International Physical Activity Questionnaires (IPAQ) comprises a set of 4 questionnaires. The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health related physical activity.
Change in Dietary Screening Questionnaire (DSQ) scores across an eight week study. | Change from baseline and then at end of study [Day 57]
  The DSQ assesses frequency of food intake, and is provided by the National Health and Nutrition Examination Survey (NHANES).
Changes in Health and Performance Questionnaire (HPQ) Question A9 scores across an eight week study. | Change from baseline and then at end of study [Day 57]
  The HPQ Question A9 is 7 items taken from the HPQ assessing work performance, with responses ranging from "All of the time" to "None of the time".
Change in the Questionnaire on Use of Evening Electronics (QUEEN) scores across an eight (8) week study | Change from baseline and then at end of study [Day 57]
  The Questionnaire on Use of Evening Electronics (QUEEN) consists of 40 items assessing the use of electronic devices at night.
Change in the Fatigue Severity Scale (FSS) across an eight (8) week study. | Change from baseline and then at end of study [Day 57]
  Fatigue Severity Scale (FSS) is a well-validated 9-item clinical measure that assesses overall levels of mental and physical fatigue, with answers ranging from 1- "Strongly Disagree" to 7-"Strongly Agree".
Change in Work Hours and Timing Questionnaire scores across an eight (8) week Study | [Time Frame: Change from baseline and then at end of study [Day 57]
  Work Hours and Timing Questionnaire (WHAT) is a 14-item questionnaire assessing employment status and work timing.
Change in Sleep Continuity questionnaire scores across an eight (8) weeks study | [Time Frame: Change from baseline and then at end of study [Day 57]
  The Sleep Continuity questionnaire consists of 15 items and assesses sleep timing and sleep difficulties during weeknights and weekdays.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States